CLINICAL TRIAL: NCT07050030
Title: Association of Preoperative Coronary Calcium Score and Postoperative Atrial Arrythmia in Patients Undergoing Robot-assisted Esophagectomy: Prospective Observational Study
Status: Not yet recruiting | Type: Observational
Sponsor: Yonsei University (Other)
Responsible Party: Sponsor
Other Study IDs: 4-2025-0388
Record Dates: First submitted 2025-06-25; First posted 2025-07-03 (Actual); Last update posted 2025-07-03 (Actual); Status verified 2025-06

CONDITIONS: Patients Undergoing Robot-assisted Esophagectomy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- patients undergoing robot-assisted esophagectomy: Adult patients aged 20 years or older and who underg robot-assisted esophagectomy

SUMMARY:
This study aimed to evaluate the relationship between coronary artery calcium score measured before surgery and the incidence of atrial fibrillation after robot-assisted esophagectomy.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged 20 years or older undergoing robotic esophagectomy
* Patients who underwent preoperative coronary computed tomography (CT) with a valid coronary artery calcium score

Exclusion Criteria:

* emergency surgery
* patients who cannot read consent forms(e.g., illiterate, foreigner, etc.)
* patients with cognitive dysfunction
* pregnant, lactating women
* history of atrial fibrillation prior to surgery

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients undergoing robotic esophagectomy
Sampling Method: Non-Probability Sample
Enrollment: 300 (Estimated)
Dates: Start 2025-07-07 (Estimated); Primary Completion 2029-07-07 (Estimated); Study Completion 2030-01-07 (Estimated)

PRIMARY OUTCOMES:
Incidence of postoperative atrial fibrillation | within 30 days postoperatively
  Incidence of postoperative atrial fibrillation within 30 days after surgery.

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Anesthesiology and Pain Medicine, Anesthesia and Pain Research Institue, Yonsei Universiy College of Medicine, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: Undecided